CLINICAL TRIAL: NCT03286257
Title: Can Exercise Training Reduce the Frequency and Severity of Hot Flushes Associated With Breast Cancer Treatment?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Principal Investigator, Helen Jones, Professor of Cardiovascular Physiology, Liverpool John Moores University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16/NW/0166
Record Dates: First submitted 2017-09-09; First posted 2017-09-18 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: Vascular function; Vascular structure; Thermoregulation; Hot flushes; Cerebral blood flow; Exercise training
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Intervention (Experimental): Participants will complete a partially supervised 4 month exercise program consisting of 3-5 sessions/week at a moderate intensity (40-75% heart rate (HR) reserve) at Liverpool Lifestyles gyms. Participants will be given free access to the Wellness Key System© when using the Lifestyles exercise equipment which allows researchers to remotely track the exercise intensity of participants accurately.
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — A partially supervised 16-week moderate intensity exercise intervention consisting of 3-5 sessions per week.

SUMMARY:
In brief, this study sets out to understand if exercise training can reduce the frequency and severity of hot flushes associated with breast cancer treatment.

DETAILED DESCRIPTION:
In detail, the aim of this research project is to investigate whether improving temperature control mechanisms including vascular function, with exercise training is beneficial in alleviating hot flushes in breast cancer patients and their associated quality of life symptoms. Participants will be recruited at least 3-months post breast cancer treatment (surgery, radio-therapy, chemotherapy). This time point has been chosen for this study to allow patients to fully engage in the exercise intervention following treatment. All participants will be asked to attend the laboratory at Liverpool John Moores University on 4 separate occasions; 2 visits pre- and 2 visits following the exercise intervention for data collection including measures of vascular health, physical activity, sedentary behaviour, and fitness. The investigators will also gain information on food intake and incidence of hot flushes across a 7-day period pre- and post the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Pre-menopausal, Peri-menopausal or post-menopausal
* >4 hot flushes per day
* Female
* Treated with tamoxifen or aromatase inhibitor

Exclusion Criteria:

* Uncontrolled or severe hypertension (blood pressure > 160/100 mm Hg)
* Any previous injury preventing exercise
* Type 1 or 2 diabetes
* Anti-depressants
* Currently undergoing chemotherapy or radiotherapy
* Current smoker
* Cannot readily read and understand English

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Thermoregulation | Change from pre- to post- 16 week exercise intervention
  Participants will wear a tube-lined suit that allows manipulation of skin temperature by heating the water passed through the tubes. Core temperature will be increased by 1 degree (monitored using a temperature pill) with sweat rate and skin temperature recordings taken at 5minute intervals across 1 hour of heating. Thermoregulation will be compared during this hour to that of the post-exercise intervention re-test.
Change in Skin Blood Flow | Change from pre- to post- 16 week exercise intervention
  The change in skin blood flow will be measured using laser Doppler probes at the forearm.

SECONDARY OUTCOMES:
Change in Cerebral Blood Flow | Change from pre- to post- 16 week exercise intervention
  Change in cerebral blood flow will be assessed using transcranial Doppler ultrasound to measure brain blood flow.
Change in Vascular Function | Change from pre- to post- 16 week exercise intervention
  Vascular function will be measured via endothelial-dependent flow mediated dilation of the brachial artery and reported as a percentage change.
Change in Vascular Structure | Change from pre- to post- 16 week exercise intervention
  Vascular structure will be measured at the carotid artery using ultrasound imaging to clearly visualise the artery. The image will be adjusted so artery wall thickness can be clearly seen with a 30 second recording taken at 3 different angles. The average of the three angles will be calculated with results reported as change in millimetres.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Jones, Study Director — Professor
Locations (1):
- Research Institute for Sport and Exercise Sciences (RISES), Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No